CLINICAL TRIAL: NCT04065763
Title: Correlation of the Dural Sac Dimension With the Spread of Spinal Anesthesia in Elderly Patients
Brief Title: Correlation of the Dural Sac Dimension With the Spread of Spinal Anesthesia
Status: Completed | Type: Observational
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, Associate professor, SMG-SNU Boramae Medical Center
Other Study IDs: 2019-02
Record Dates: First submitted 2019-08-12; First posted 2019-08-22 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Elderly Patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ultrasound assessment of dural sac dimension — Dural sac dimension is assessed using ultrasonography in the lateral decubitus position for spinal anesthesia.

SUMMARY:
Cerebrospinal fluid volume is an important factor that influences peak block height and regression of sensory and motor blockade. The aim of this study is to evaluate the effect of dural sac dimension on the spread of spinal anesthesia in elderly patient using ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for elective surgery under spinal anesthesia

Exclusion Criteria:

* Known anatomical abnormality or pathology in the spine
* History of lumbar spinal surgery or compression fracture
* Height less than 150 cm

Min Age: 65 Years | Sex: Female
Age Groups: Older Adult
Study Population: Female patients older than 65 years of age who are undergoing elective surgery under spinal anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-14 (Actual)

PRIMARY OUTCOMES:
Correlation between the dural sac dimension and spinal anesthesia spread (peak sensory block) | At 30 minutes after the induction of spinal anesthesia
  The dural sac dimension is assessed before spinal anesthesia. After spinal anesthesia, the sensory and motor level are evaluated. Then, the correlation between the dural sac dimension and spinal anesthesia blockade is assessed.

SECONDARY OUTCOMES:
Correlation between the dural sac dimension and duration of spinal anesthesia | At 30 minutes after the end of surgery
  The sensory and motor regression are assessed. Then, the correlation between the dural sac dimension and the duration of spinal blockade is assessed.
Correlation between the dural sac dimension and body mass index | 5 minutes before spinal anesthesia
  Correlation between the dural sac dimension and body mass index is assessed.
Correlation between the dural sac dimension and waist circumference | 5 minutes before spinal anesthesia
  Correlation between the dural sac dimension and waist circumference is assessed.
Correlation between the dural sac dimension and age | 5 minutes before spinal anesthesia
  Correlation between the dural sac dimension and age is assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- SMG-SNU Boramae Medical Center, Seoul, South Korea